CLINICAL TRIAL: NCT06136143
Title: Double-blind Randomized Controlled Clinical Study of the Predictability of Using Plenum® Osshp in Maxillary Sinus Elevation Surgery
Brief Title: Plenum® Osshp in Maxillary Sinus Elevation Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: M3 Health (Industry)
Collaborators: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Plenum Oss 001
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Oral Surgical Procedures
Keywords: Maxillary Sinus; Synthetic Bone Graft; Autogenous Bone Graft; Platelet Rich Fibrin
MeSH Terms: interventions — Sinus Floor Augmentation; proliferation regulatory factors, human urine

STUDY DESIGN:
Intervention Model Description: For this, forty (40) participants will be recruited for procedure surgery of maxillary sinus elevation and subsequent installation of dental implants after 06 months of postoperative. And then, the participants will divided into 4 groups, which will have 10 participants each, namely: Group 1: Autogenous bone; Group 2: Plenum® Osshp; Group 3: Plenum® Osshp; + i-PRF and Group 4: Plenum® Osshp; + autogenous bone. To evaluate the primary outcome, volumetric analysis will be performed by obtaining computed tomography scans at 15 days (T1) and 6 months (T2) after graft surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Autogenous bone graft (Active Comparator): The maxillary sinus will treated with autogenous bone graft.
  Interventions: Procedure: Group 1: Autogenous bone graft
- Group 2: Plenum® Osshp (Experimental): The maxillary sinus will treated with Plenum® Osshp.
  Interventions: Procedure: Group 2: Plenum® Osshp
- Group 3: Plenum® Osshp; + i-PRF (Experimental): The maxillary sinus will treated with Plenum® Osshp associated with i-PRF (i-PR - injectable platelet-rich fibrin).
  Interventions: Procedure: Group 3: Plenum® Osshp; + i-PRF
- Group 4: Plenum® Osshp + autogenous bone graft (Experimental): The maxillary sinus will treated with Plenum® Osshp associated with autogenous bone graft.
  Interventions: Procedure: Group 4: Plenum® Osshp + autogenous bone graft

INTERVENTIONS:
Procedure: Group 1: Autogenous bone graft — The maxillary sinus will be grafted with the autogenous bone graft.
  Other Names: Maxillary sinus elevation surgery; Maxillary sinus augmentation; Maxillary sinus lift
  Arms: Group 1: Autogenous bone graft
Procedure: Group 2: Plenum® Osshp — The maxillary sinus will be grafted with the Plenum Oss hp (Plenum, Brazil) medical device.
  Other Names: Maxillary sinus elevation surgery; Maxillary sinus augmentation; Maxillary sinus lift
  Arms: Group 2: Plenum® Osshp
Procedure: Group 3: Plenum® Osshp; + i-PRF — The maxillary sinus will be grafted with the Plenum Oss hp (Plenum, Brazil) medical device associated with i-PRF.
  Other Names: Maxillary sinus elevation surgery; Maxillary sinus augmentation; Maxillary sinus lift
  Arms: Group 3: Plenum® Osshp; + i-PRF
Procedure: Group 4: Plenum® Osshp + autogenous bone graft — The maxillary sinus will be grafted with the Plenum Oss hp (Plenum, Brazil) medical device associated with autogenous bone graft.
  Other Names: Maxillary sinus elevation surgery; Maxillary sinus augmentation; Maxillary sinus lift
  Arms: Group 4: Plenum® Osshp + autogenous bone graft

SUMMARY:
The aim of this study is to qualitatively and quantitatively evaluate bone neoformation in maxillary sinus lift surgery filled with Plenum® Oss hp, compared to filling with autogenous bone, and to verify the association of Plenum® Osshp with i-PRF (i-PR - injectable platelet-rich fibrin). For this, forty (40) participants will be recruited, divided into 4 groups, which will have 10 participants each, namely: Group 1: Autogenous bone; Group 2: Plenum® Osshp; Group 3: Plenum® Osshp; + i-PRF and Group 4: Plenum® Osshp; + autogenous bone. To evaluate the primary outcome, volumetric analysis will be performed by obtaining computed tomography scans at 15 days (T1) and 6 months (T2) after graft surgery, with the aid of a volumetric tomography machine for dentofacial images. The values obtained at T2 will be subtracted from those obtained from T1 to obtain the volumetric stability value. After six months of repair, biopsies will be performed using a trephine drill, followed by the installation of implants and healers. Through microcomputed tomography analysis, the parameters of bone volume fraction (BV/TV), total porosity (Po.Tot), trabecular thickness (Tb.Th), number of trabeculae (Tb.N) and separation of trabeculae (Tb.Sp) will be evaluated. Histomorphometric analysis will be performed to obtain the areas of bone neoformation, connective tissue and remaining biomaterial that will be calculated for each area of the sample (cervical, intermediate, and apical) and later summed, obtaining the total representative area of the sample. Through immunohistochemical analysis, specific primary antibodies to Runx2, VEGF, Osteocalcin (OC) and Tartrate-Resistant Acid Phosphatase (TRAP) will be identified. The occurrence of adverse events will be collected through the analysis of pain, infection, and edema. The quantitative results of the histomorphometric, microtomographic, and volumetric stability analysis will be tabulated and submitted to the ANOVA test, and if they present a statistically significant difference, it will be followed by the Tukey test (post hoc). A significance level of p<0.05 will be adopted for all tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with alveolar ridge atrophy, with bone remnant less than 5 mm in height, with adequate bone volume in the ramus and/or symphysis region;
* Over 18 years old;
* And that they have signed the informed consent form.

Exclusion Criteria:

* Smokers;
* Patients with uncontrolled systemic diseases;
* Patients with blood dyscrasias;
* Patients with sinus pathologies;
* Patients who take or have used medications that interfere with bone turnover;
* Patients irradiated in the head and neck region;
* Pregnant patients;
* Patients with untreated periodontal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Rate of the maintenance of volume in the maxillary sinus region. | Fifteen days (T1) and six months (T2) from postoperative.
  Computed tomography scans were performed and compared after graft surgery (T1) and after 6 months of repair (T2). The maintenance of the volume will be defined by the difference in the area of T2-T1.

SECONDARY OUTCOMES:
Rate of the bone neoformation of the synthetic graft in comparison with the autogenous graft and in association with i-PRF. | Six months from postoperative.
  Microcomputed tomography analysis using the following variables: Bone volume fraction, total porosity, trabecular thickness, number of trabeculae and separation of trabeculae.
Rate of the areas of bone neoformation, connective tissue and remnant synthetic graft. | Six months from postoperative.
  Histomorphometric analysis of the experimental groups.
Rate of influence of the use of synthetic grafts on newly formed bone tissue, in comparison with autogenous grafts and in association with i-PRF. | Six months from postoperative.
  Quantification of specific marker for Runx2.
Rate of influence of the use of synthetic grafts on newly formed bone tissue, in comparison with autogenous grafts and in association with i-PRF. | Six months from postoperative.
  Quantification of specific marker for VEGF.
Rate of influence of the use of synthetic grafts on newly formed bone tissue, in comparison with autogenous grafts and in association with i-PRF. | Six months from postoperative.
  Quantification of specific marker for Osteocalcin (OC)
Rate of influence of the use of synthetic grafts on newly formed bone tissue, in comparison with autogenous grafts and in association with i-PRF. | Six months from postoperative.
  Quantification of specific marker for Tartrate-Resistant Acid Phosphatase (TRAP).

CONTACTS AND LOCATIONS:
Overall Officials: Sybele Specian, PhD, Study Director — Plenum (M3 Health)
Locations (1):
- Universidade Estadual Paulista - UNESP, Araraquara, São Paulo, Brazil